CLINICAL TRIAL: NCT07264842
Title: Triple Antibiotic Paste Versus Simvastatin for LSTR Treatment of Primary Molars With Pulp Necrosis: A Randomized Controlled Trial
Brief Title: Triple Antibiotic Paste vs Simvastatin for Lesion Sterilization and Tissue Repair in Primary Molars.
Acronym: LSTR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Waleed Mumtaz, Postgraduate Trainee- FCPS, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3379/DUHS//Approval/2024/175
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Pulpal Necrosis
Keywords: Lesion Sterilization and Tissue Repair
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Wound Healing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simvastatin (Experimental): Lesion Sterilization and Tissue Repair using Simvastatin.
  Interventions: Combination Product: Lesion Sterilization and Tissue Repair
- Triple Antibiotic Paste (Active Comparator): Lesion Sterilization and Tissue Repair using triple antibiotic paste
  Interventions: Combination Product: Lesion Sterilization and Tissue Repair

INTERVENTIONS:
Combination Product: Lesion Sterilization and Tissue Repair — Lesion sterilization and Tissue Repair includes removal of any debris from the pulp chamber of the primary tooth and filling with triple antibiotic paste or simvastatin followed by sealed with the restoration.

SUMMARY:
This randomized, double-blinded, parallel-controlled clinical trial aims to compare the effectiveness of Triple Antibiotic Paste (TAP) and Simvastatin in Lesion Sterilization and Tissue Repair (LSTR) of primary molars with pulp necrosis.

A total of 60 children (aged 5-8 years) with non-vital primary molars will be recruited from the Department of Operative Dentistry and Endodontics, Dow International Dental College, Karachi. Participants will be randomly assigned to one of two groups:

Group 1 (Control): LSTR using Triple Antibiotic Paste (Ciprofloxacin + Metronidazole + Cefixime).

Group 2 (Intervention): LSTR using Simvastatin paste.

Both materials will be placed after non-instrumentation cleaning and sealed with glass ionomer cement, followed by stainless steel crown placement. Patients will be evaluated clinically and radiographically at 1, 2, and 3 months post-treatment.

Primary outcomes include clinical success (absence of pain, swelling, or sinus tract) and radiographic success (reduction or absence of periapical radiolucency). Data will be analyzed using SPSS v26, with chi-square and t-tests applied as appropriate; p < 0.05 will be considered significant.

This study seeks to determine whether Simvastatin, owing to its antibacterial, anti-inflammatory, and regenerative properties, can serve as a viable alternative to antibiotic-based LSTR in managing necrotic primary teeth.

ELIGIBILITY:
Inclusion Criteria:

* Young, healthy patient, ranging in age from 5-8 years.
* Has parents/ guardians who give consent to allow their minor to participate in the study and willing to monitor their progress.
* Having maxillary and mandibular primary molars with:

  * Spontaneous pain or tenderness to percussion.
  * Deep cavity extending to the pulp chamber.
  * Chronic Abscess or draining sinus.
  * Restorable.
  * To be kept for less than a year.
  * Irregular mobility that is not related to exfoliation.

Exclusion Criteria:

* Uncooperative patients.
* Children with a history of allergic reaction with antibiotics.
* Teeth with physiological root resorption but root length is more than two thirds, root canal obliteration, severe internal resorption, internal calcifications, or piercing into the bifurcation.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 1 month, 2 month and 3 month.
  Reduction or absence in pain and swelling will be considered as clinical success.
Radiographic Success | 1 month, 2 month and 3 month
  Reduction or absence of radiolucency will be considered as radiographic success.

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Dr. Farah Naz Biyabani, FCPS, Study Director — Dow University of Health Sciences
Locations (1):
- Dow International Dental College, Chanesar goth., Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided